CLINICAL TRIAL: NCT07131241
Title: Research on Dynamic Risk Prediction for Patients With Pulmonary Hypertension Based on Multimodal Data Fusion: A Prospective Observational Study
Brief Title: PH-DyPred: A Multimodal Dynamic Risk Prediction Study in Pulmonary Hypertension
Acronym: PH-DyPred
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Dajun Chai, Professor and Chief Physician, Department of Cardiology, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MRCTA,ECFAH of FMU[2025]716
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Dynamic Risk Prediction; Multimodal Data Fusion; Echocardiography; Right Heart Function; Cardiac Magnetic Resonance
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, urine, and stool samples will be collected and stored for future analysis. Blood-derived samples will be used for genomic, proteomic, metabolomic, and microRNA profiling. Urine samples will be analyzed for renal biomarkers and metabolomic profiling. Stool samples will be used for microbiome analysis. All specimens will be processed and stored according to standardized protocols in a secure biobank. Biospecimens are linked to clinical, imaging, and follow-up data via de-identified subject codes for integrated analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected PH by Echocardiography: This study includes a prospective observational cohort of patients with suspected pulmonary hypertension (PH), identified by transthoracic echocardiography (TTE) showing a pulmonary artery systolic pressure (PASP) ≥35 mmHg. No experimental intervention will be applied. Participants will undergo comprehensive data collection, including echocardiography, cardiac magnetic resonance imaging (CMR), electrocardiography (ECG), laboratory testing, and biospecimen sampling (blood, urine, and stool). Follow-up will occur every 6 months for up to 3 years to record clinical outcomes and support the development of a dynamic, multimodal risk prediction model based on artificial intelligence.

SUMMARY:
Pulmonary hypertension (PH) is a progressive cardiopulmonary disease characterized by elevated pulmonary artery pressure and vascular remodeling, which leads to right heart failure and increased mortality. Despite advances in diagnostics, risk stratification remains limited due to the disease's heterogeneity. This study aims to develop and validate a dynamic risk prediction model for PH by integrating multimodal data-including echocardiography, Cardiac MRI, PET-MR, ECG, biomarkers, and clinical features-using advanced machine learning algorithms. The study will establish a prospective cohort of PH patients to explore predictive markers, stratify prognosis, and provide a scientific basis for early warning and individualized management.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study designed to investigate dynamic risk prediction in patients diagnosed with pulmonary hypertension (PH). The study will collect multimodal clinical data-comprising imaging (echocardiography, cardiac MRI, PET-MR), electrocardiographic parameters, blood-based biomarkers, and demographic and clinical information-at baseline and follow-up intervals. The core objective is to develop a data fusion-based prognostic model capable of predicting adverse outcomes such as hospitalization, functional deterioration, or mortality. Machine learning methods will be employed to identify key predictive features. The model will be validated internally and externally across different subgroups. The study seeks to inform individualized risk-based decision-making and advance precision screening in PH care.

In addition, biospecimens will be collected to support comprehensive multi-omics profiling. Whole blood, serum, plasma, urine, and stool samples will be obtained and processed using standardized protocols. Blood-derived samples will be used for genomic, proteomic, metabolomic, and microRNA analyses; urine specimens will support metabolomic and renal biomarker assays; and stool samples will be used for gut microbiome sequencing. All biospecimens will be stored in a secure biobank and linked with clinical, imaging, and longitudinal follow-up data using de-identified subject codes to enable integrated multimodal analyses and facilitate future exploratory investigations of disease mechanisms and biomarker discovery.

Health economic evaluation, including cost-effectiveness and budget impact analyses, will be conducted using collected data on healthcare resource utilization, direct medical costs, and clinical outcomes to inform future policy and reimbursement decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Pulmonary artery systolic pressure (PASP) ≥35 mmHg as estimated by echocardiography
* Provided written informed consent

Exclusion Criteria:

* Severe hepatic or renal insufficiency
* Malignancy under active treatment
* Severe infection
* Active autoimmune disease
* Major surgery within the past 3 months
* Pregnant or breastfeeding women
* Severe psychiatric disorder impairing ability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years) undergoing transthoracic echocardiography. Participants with a pulmonary artery systolic pressure (PASP) ≥35 mmHg on echocardiography will be included as suspected pulmonary hypertension cases. This cohort represents a real-world population at risk for or with early-stage pulmonary hypertension, suitable for developing dynamic risk prediction models based on multimodal data integration.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical worsening | Up to 36 months
  Defined as any of the following: hospitalization for PH, escalation of therapy, 6MWD decrease >15%, WHO-FC worsening, or death. Measured from baseline.
All-cause mortality | Up to 36 months
  Death from any cause during follow-up, as confirmed by medical records or death registry.

SECONDARY OUTCOMES:
Composite risk score performance (AUC) | At baseline and follow-up every 6 months
  Area under the ROC curve for the multimodal model predicting adverse outcomes.
Changes in NT-proBNP levels | Baseline, 6, 12, 24, 36 months
  Evaluate biomarker dynamics and predictive value.
Hospitalization rate for PH-related causes | Up to 36 months
  Frequency of hospital admissions due to PH complications.
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) Measured by Transthoracic Echocardiography | Baseline, 6, 12, 24, 36 months
  TAPSE (mm) will be measured via transthoracic echocardiography to evaluate longitudinal right ventricular systolic function over time.
Change in Right Ventricular Diameter Measured by Transthoracic Echocardiography | Baseline, 6, 12, 24, 36 months
  Right ventricular internal diameter (mm) will be assessed by echocardiography as an indicator of RV structural remodeling.
Change in Right Ventricular Fractional Area Change (RVFAC) Measured by Transthoracic Echocardiography | Baseline, 6, 12, 24, 36 months
  RVFAC (%) will be calculated as the percentage change in RV area between end-diastole and end-systole to assess systolic function.
Change in Right Ventricular Ejection Fraction (RVEF) Measured by Cardiac Magnetic Resonance Imaging | Baseline, 6, 12, 24, 36 months
  RVEF (%) will be quantified using cardiac magnetic resonance imaging to evaluate global systolic function.
Change in Right Ventricular End-Diastolic Volume Measured by Cardiac Magnetic Resonance Imaging | Baseline, 6, 12, 24, 36 months
  Right ventricular end-diastolic volume (mL) will be measured by CMR to assess structural remodeling over time.
Change in Right Ventricular Mass Measured by Cardiac Magnetic Resonance Imaging | Baseline, 6, 12, 24, 36 months
  Right ventricular mass (grams) will be measured by CMR as an index of ventricular hypertrophy and remodeling.
Change in Right Ventricular FAPI Uptake (SUVmean) Measured by FAPI PET-MR | Baseline, 12, 24, and 36 months
  tandardized uptake value mean (SUVmean) of FAPI in the right ventricular free wall will be quantified using PET-MR imaging to assess fibroblast activation and myocardial fibrotic activity over time in patients with pulmonary hypertension.
Change in Right Ventricular FAPI Uptake (SUVmax) Measured by FAPI PET-MR | Baseline, 12, 24, and 36 months
  Maximum standardized uptake value (SUVmax) of FAPI in the right ventricle will be measured via PET-MR as an indicator of peak regional fibroblast activation.
Change in Right Ventricular FAPI Uptake Ratio Relative to Left Ventricle (SUVratio) Measured by FAPI PET-MR | Baseline, 12, 24, and 36 months
  The ratio of right ventricular to left ventricular myocardial FAPI uptake (SUVmean RV/SUVmean LV) will be calculated as a normalized index of right ventricular fibrotic remodeling.

OTHER OUTCOMES:
Longitudinal changes in health-related quality of life (HRQoL) among patients with suspected or confirmed pulmonary hypertension | Baseline, 6, 12, 24, and 36 months
  Health-related quality of life (HRQoL) will be assessed using validated instruments such as the EQ-5D-3L and/or the emPHasis-10 questionnaire, both commonly used in pulmonary hypertension research. The emPHasis-10 is a disease-specific, patient-reported outcome measure developed for individuals with pulmonary hypertension, covering domains such as breathlessness, fatigue, social limitation, and psychological burden. Changes in HRQoL scores will be evaluated over time and correlated with clinical events (e.g., hospitalization, WHO functional class deterioration), imaging parameters (e.g., RV function), biomarkers (e.g., NT-proBNP), and model-predicted risk strata. Analyses will include repeated measures ANOVA or mixed-effects modeling to examine within-subject longitudinal chan
Area Under the ROC Curve (AUC) of the Multimodal Risk Prediction Model | Baseline, 12, 24, 36 months
  The area under the receiver operating characteristic curve (AUC) will be calculated to evaluate the discrimination performance of the multimodal dynamic risk prediction model for adverse outcomes.
Harrell's Concordance Index (C-index) of the Multimodal Risk Prediction Model | Baseline, 12, 24, 36 months
  The concordance index (C-index) will be computed to assess the predictive accuracy of the multimodal risk prediction model.
Calibration Slope of the Multimodal Risk Prediction Model | Baseline, 12, 24, 36 months
  Calibration slope will be estimated to measure agreement between predicted and observed risks in the dynamic risk prediction model.
Net Benefit Derived from Decision Curve Analysis of the Multimodal Risk Prediction Model | Baseline, 12, 24, 36 months
  Net benefit will be calculated using decision curve analysis to evaluate the clinical usefulness of the multimodal risk prediction model in guiding clinical decision-making.
Correlation between NT-proBNP Concentration (pg/mL) and Right Ventricular Ejection Fraction (RVEF) | Baseline, 6, 12, 24, and 36 months
  NT-proBNP concentration will be measured in plasma using a standardized immunoassay (pg/mL). Pearson correlation coefficients (r) will be calculated between NT-proBNP levels and right ventricular ejection fraction (RVEF, %) measured by cardiac MRI.
  Unit of Measure: Correlation coefficient (r)
Correlation between NT-proBNP Concentration (pg/mL) and Right Ventricular End-Diastolic Volume (RVEDV) | Baseline, 6, 12, 24, and 36 months
  NT-proBNP concentration measured by immunoassay (pg/mL) will be correlated with right ventricular end-diastolic volume (mL) assessed by cardiac MRI. Pearson correlation coefficients (r) will be calculated at each follow-up time point.
  Unit of Measure: Correlation coefficient (r)
Correlation between NT-proBNP Concentration (pg/mL) and TAPSE | Baseline, 6, 12, 24, and 36 months
  NT-proBNP levels (pg/mL) obtained by immunoassay will be correlated with tricuspid annular plane systolic excursion (TAPSE, mm) measured on transthoracic echocardiography using Pearson correlation.
  Unit of Measure: Correlation coefficient (r)
Correlation between NT-proBNP Concentration (pg/mL) and Right Ventricular Longitudinal Strain | Baseline, 6, 12, 24, and 36 months
  NT-proBNP values (pg/mL) will be correlated with right ventricular longitudinal strain (%) measured by speckle-tracking echocardiography. Pearson correlation coefficients (r) will be reported.
  Unit of Measure: Correlation coefficient (r)
Correlation between NT-proBNP Concentration (pg/mL) and Right Ventricular Fractional Area Change (RVFAC) | Baseline, 6, 12, 24, and 36 months
  Plasma NT-proBNP level (pg/mL) will be correlated with right ventricular fractional area change (RVFAC, %) measured using echocardiography, and correlation coefficients (r) will be calculated over time.
  Unit of Measure: Correlation coefficient (r)
Association between Baseline NT-proBNP Concentration and Time to Clinical Worsening | Up to 36 months
  Baseline plasma NT-proBNP levels (pg/mL), measured using a standardized immunoassay, will be analyzed using Cox proportional hazards models to assess their association with time to clinical worsening, defined as hospitalization for pulmonary hypertension, WHO functional class deterioration, or death.
  Unit of Measure: Hazard ratio (HR)
Association between Baseline NT-proBNP Concentration and Model-Predicted Risk Categories | Baseline, 6, 12, 24, and 36 months
  Baseline NT-proBNP concentration (pg/mL), measured using a standardized immunoassay, will be analyzed using multinomial or logistic regression models to evaluate its association with model-predicted risk categories (e.g., low-, intermediate-, and high-risk strata) generated by the multimodal dynamic risk prediction model.
  Unit of Measure: Odds ratio (OR)

CONTACTS AND LOCATIONS:
Overall Officials: Dajun Chai, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including demographic information, clinical characteristics, imaging parameters (echocardiography and CMR), ECG data, laboratory test results, biospecimen profiles (e.g., biomarkers, multi-omics), and follow-up outcomes, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available beginning 24 months after the primary study completion date and remain accessible for up to 24 months.
Access Criteria: Qualified researchers with a scientifically sound proposal may request access to the data. Requests will be evaluated by the study steering committee. Approved users must sign a data use agreement ensuring compliance with privacy, ethical, and scientific standards.
URL: https://www.fjmu.edu.cn

REFERENCES:
- [Background] Fauvel C, Gomberg-Maitland M, Benza RL. Risk Stratification in Pulmonary Hypertension: We Need to "GoDeeper"! Chest. 2024 Sep;166(3):420-422. doi: 10.1016/j.chest.2024.05.020. No abstract available. PMID 39260943
- [Background] Lorenzatti D, Motwani M. Cardiovascular magnetic resonance in pulmonary hypertension: Keeping it simple. Prog Cardiovasc Dis. 2025 May-Jun;90:116-118. doi: 10.1016/j.pcad.2025.04.010. Epub 2025 Apr 26. No abstract available. PMID 40294712
- [Background] Kjellstrom B, Lindholm A, Ostenfeld E. Cardiac Magnetic Resonance Imaging in Pulmonary Arterial Hypertension: Ready for Clinical Practice and Guidelines? Curr Heart Fail Rep. 2020 Oct;17(5):181-191. doi: 10.1007/s11897-020-00479-7. PMID 32870447
- [Background] Meyer GMB, Spilimbergo FB, Altmayer S, Pacini GS, Zanon M, Watte G, Marchiori E, Hochhegger B. Multiparametric Magnetic Resonance Imaging in the Assessment of Pulmonary Hypertension: Initial Experience of a One-Stop Study. Lung. 2018 Apr;196(2):165-171. doi: 10.1007/s00408-018-0097-7. Epub 2018 Feb 12. PMID 29435739
- [Background] van de Veerdonk MC, Kind T, Marcus JT, Mauritz GJ, Heymans MW, Bogaard HJ, Boonstra A, Marques KM, Westerhof N, Vonk-Noordegraaf A. Progressive right ventricular dysfunction in patients with pulmonary arterial hypertension responding to therapy. J Am Coll Cardiol. 2011 Dec 6;58(24):2511-9. doi: 10.1016/j.jacc.2011.06.068. PMID 22133851
- [Background] Small M, Perchenet L, Bennett A, Linder J. The diagnostic journey of pulmonary arterial hypertension patients: results from a multinational real-world survey. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666231218886. doi: 10.1177/17534666231218886. PMID 38357903
- [Background] Hameed A, Condliffe R, Swift AJ, Alabed S, Kiely DG, Charalampopoulos A. Assessment of Right Ventricular Function-a State of the Art. Curr Heart Fail Rep. 2023 Jun;20(3):194-207. doi: 10.1007/s11897-023-00600-6. Epub 2023 Jun 5. PMID 37271771
- [Background] Rachedi NS, Tang Y, Tai YY, Zhao J, Chauvet C, Grynblat J, Akoumia KKF, Estephan L, Torrino S, Sbai C, Ait-Mouffok A, Latoche JD, Al Aaraj Y, Brau F, Abelanet S, Clavel S, Zhang Y, Guillermier C, Kumar NVG, Tavakoli S, Mercier O, Risbano MG, Yao ZK, Yang G, Ouerfelli O, Lewis JS, Montani D, Humbert M, Steinhauser ML, Anderson CJ, Oldham WM, Perros F, Bertero T, Chan SY. Dietary intake and glutamine-serine metabolism control pathologic vascular stiffness. Cell Metab. 2024 Jun 4;36(6):1335-1350.e8. doi: 10.1016/j.cmet.2024.04.010. Epub 2024 May 2. PMID 38701775
- [Background] Yorke J, Corris P, Gaine S, Gibbs JS, Kiely DG, Harries C, Pollock V, Armstrong I. emPHasis-10: development of a health-related quality of life measure in pulmonary hypertension. Eur Respir J. 2014 Apr;43(4):1106-13. doi: 10.1183/09031936.00127113. Epub 2013 Nov 14. PMID 24232702
- [Background] Zhao W, Huang Z, Diao X, Yang Z, Zhao Z, Xia Y, Zhao Q, Sun Z, Xi Q, Huo Y, Xu O, Geng J, Li X, Duan A, Zhang S, Gao L, Wang Y, Li S, Luo Q, Liu Z. Development and validation of multimodal deep learning algorithms for detecting pulmonary hypertension. NPJ Digit Med. 2025 Apr 10;8(1):198. doi: 10.1038/s41746-025-01593-3. PMID 40205021
- [Background] Rich S, Haworth SG, Hassoun PM, Yacoub MH. Pulmonary hypertension: the unaddressed global health burden. Lancet Respir Med. 2018 Aug;6(8):577-579. doi: 10.1016/S2213-2600(18)30268-6. Epub 2018 Jun 29. No abstract available. PMID 30072105
- [Background] Humbert M, Kovacs G, Hoeper MM, Badagliacca R, Berger RMF, Brida M, Carlsen J, Coats AJS, Escribano-Subias P, Ferrari P, Ferreira DS, Ghofrani HA, Giannakoulas G, Kiely DG, Mayer E, Meszaros G, Nagavci B, Olsson KM, Pepke-Zaba J, Quint JK, Radegran G, Simonneau G, Sitbon O, Tonia T, Toshner M, Vachiery JL, Vonk Noordegraaf A, Delcroix M, Rosenkranz S; ESC/ERS Scientific Document Group. 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Heart J. 2022 Oct 11;43(38):3618-3731. doi: 10.1093/eurheartj/ehac237. No abstract available. PMID 36017548
- See also: Description: Official website of the First Affiliated Hospital of Fujian Medical University, the lead institution responsible for this study. The site includes institutional information, clinical departments, research governance, and contact information. — https://www.fjmu.edu.cn
- Available data/document: Individual Participant Data Set — https://www.fjmu.edu.cn — For more information, please contact: dajunchai@126.com